CLINICAL TRIAL: NCT01987167
Title: Potential Neuroprotection With ACTHAR Following Acute Optic Neuritis
Brief Title: Defining the Functional and Neuro-Protective Potential of ACTHAR in Acute Optic Neuritis
Acronym: ACHTAR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Neuro-Ophthalmologic Associates, PC (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-330; ACTHAR (Other: Questcor Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-11-06; First posted 2013-11-19 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Optic Neuritis
Keywords: acute optic neuritis
MeSH Terms: conditions — Optic Neuritis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- -ACHTHAR (Experimental): Subcutaneous ACTHAR 5 days of 80 IU and 10 Days of 40 IU
  Interventions: Drug: ACTHAR

INTERVENTIONS:
Drug: ACTHAR — Injectable Gel
  Other Names: Repository Corticotropin

SUMMARY:
The goal of the study is to determine the earliest structural changes in the optic nerve during the acute event and during the twelve months of recovery following Acthar treatment.

DETAILED DESCRIPTION:
Determine the earliest structural changes in the optic nerve during the acute event and during the twelve months of recovery following Acthar treatment.

ELIGIBILITY:
Inclusion Criteria:

* unilateral acute demyelinating optic neuritis
* Able to provide informed consent
* age 18 or older
* can perform the above listed electrophysiologic diagnostic testing
* can perform high and low contrast visual acuity and visual field perimetry

Exclusion Criteria:

* prior diagnosis of remitting/relapsing multiple sclerosis(RRMS)
* secondary progressive MS(SPMS)
* primary progressive MS (PPMS)
* undergoing treatment with medications approve for treatment of RRMS(except corticosteroids for a condition not involving central nervous system demyelination)
* prior diagnosis of systemic lupus erythematosis
* mixed connective tissue disease
* vasculitis
* sarcoidosis
* neuro-myelitis optica

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Neuro-protection | 12 months
  Functional with low contrast visual acuity in bothe the eye acutely affected by optic neuritis and the clinically unaffected eye.

SECONDARY OUTCOMES:
Preservation of retinal nerve fiber layer. | 12 months
  To define the objective (micron thickness, volumetric analysis) and subjective (histopathological changes) of spectral domain optical coherence tomography (SD-OCT) at the time of clinical presentation of acute optic neuritis and during 6 months of recovery following ACTHAR treatment.

OTHER OUTCOMES:
Preservation and/or restoration of electrophysiological parameters for patients with acute optic neuritis. | 12 months
  To define the electrophysiological changes at the onset and following an acute event of optic neuritis with Multifocal electroretinography(mERG) and visual evoked potentials (VEP)
Structural, Physiological and Metabolic changes during an acute event of optic neuritis | 12 months
  to determine the earliest structural, physiological, and metabolic changes in the optic nerve during an acute event of demyelinating optic neuritis and the natural history of these changes over 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Sergott, M.D., Principal Investigator
Locations (1):
- Neuro Ophthalmology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moster ML, Sergott RC, Leiby BE. Dalfampridine Treatment in Nonarteritic Anterior Ischemic Optic Neuropathy. J Neuroophthalmol. 2017 Sep;37(3):348-349. doi: 10.1097/WNO.0000000000000523. No abstract available. PMID 28538037